CLINICAL TRIAL: NCT07270783
Title: A Randomized, Double-Blind, Placebo-Controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of D-2570 Tablets in Healthy Subjects
Brief Title: Healthy Volunteer Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: D2570-103
Record Dates: First submitted 2025-11-12; First posted 2025-12-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 D-2570/Placebo (Experimental)
  Interventions: Drug: D-2570; Drug: Placebo
- Cohort 2 D-2570/Placebo (Experimental)
  Interventions: Drug: D-2570; Drug: Placebo
- Cohort 3 D-2570/Placebo (Experimental)
  Interventions: Drug: D-2570; Drug: Placebo

INTERVENTIONS:
Drug: D-2570 — D-2570
Drug: Placebo — Placebo

SUMMARY:
Double Blinded Healthy Volunteer study evaluating D-2570 against placebo in various doses.

DETAILED DESCRIPTION:
Double blind study evaluating the safety, tolerability and PK data of D-2570/placebo in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer subjects meeting eligibility criteria

Exclusion Criteria:

* Subjects with ongoing or history of disease or co-morbidities as assessed by Principal Investigator which would make them ineligible for the study
* Subjects with a history of drug and alcohol abuse
* Subjects taking medications, over the counter or herbal remedies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From Informed Consent through study completion, an average of 48 days
  Incidence of adverse events
Result of Pharmacokinetic endpoint | From Randomization through study completion, an average of 20 days
  Tmax
Result of Pharmacokinetic endpoint | From Randomization through study completion, an average of 20 days
  Cmax
Result of Pharmacokinetic endpoint | From Randomization through study completion, an average of 20 days
  t1/2
Result of Pharmacokinetic endpoint | From Randomization through study completion, an average of 20 days
  MRT
Result of Pharmacokinetic endpoint | From Randomization through study completion, an average of 20 days.
  AUC0-∞
Result of Pharmacokinetic endpoint | From Randomization through study completion, an average of 20 days
  AUC0-t
Result of Pharmacokinetic endpoint | From Randomization through study completion, an average of 20 days
  CL/F
Result of Pharmacokinetic endpoint | From Randomization through study completion, an average of 20 days
  Vz/F

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No